CLINICAL TRIAL: NCT01490645
Title: ProAcor: Prospective Structured Care In Acute Coronary Syndrome Registry
Brief Title: A NIS Registry of the Prospective Structured Care In Acute Coronary Syndrome
Acronym: ProAcor
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CDE-XXX-2011/1; NIS-CDE-XXX-2011/1
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS patients participating in a SCP; QoL after ACS; ASC Patients's needs
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- one group (all patients)

SUMMARY:
The purpose of the study is to analyse patient's acceptance and willingness to participate in a Structured Care Program (SCP) over 12 months following hospital discharge after Acute Coronary Syndrome (ACS) index event.

DETAILED DESCRIPTION:
ProAcor: Prospective Structured Care In Acute Coronary Syndrome Registry

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized because of ACS (ST segment elevation myocardial infarction (STEMI)), non-ST elevation myocardial infarction (NSTEMI) Unstable Angina (UA)) and planned to be discharged alive soon.

Exclusion Criteria:

* Myocardial infarction (UA, STEMI and NSTEMI) precipitated by or as a complication of surgery, trauma, or Gastrointestinal Bleeding or post- percutaneous coronary intervention (PCI).
* Myocardial infarction (UA, STEMI and NSTEMI) occurring in patients already hospitalized for other reasons.
* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, known diagnosed psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Regional centres / hospitals with a significant number of ACS patients
Sampling Method: Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The number of patients who can be guided through the structured outpatient care program offered within this project by assessing the percentage of patients with diagnosis of Acute Coronary Syndrome (ACS) following the care program. | up to 24 months
  after collecting all Case Record Form

SECONDARY OUTCOMES:
Description of reasons of premature withdrawal from the program. | up to 12 months
  after collecting all Case Record Form
Description of changes in quality of life (QoL) during the period of 12 months. | up to 12 months
  after collecting all Case Record Form
Description of acceptance of the program between subgroups (e.g. gender, risk scores, types of ACS, multimorbidity, medical treatment, therapy). | up to 12 months
  after collecting all Case Record Form
Description of patients's needs in long term care of ACS. | up to 12 months
  after collecting all Case Record Form
Description of adherence to guideline conform treatment and patients' compliance with the lifestyle changes recommended by the physician (e.g. body weight, blood pressure, Low Density Lipoprotein (LDL)). | up to 12 months
  after collecting all Case Record Form
Description of newly occurred cardiac symptoms (e.g. troponin, LVH), as determined by routine examinations by the cardiologists, which cause a declining state of health. | up to 12 months
  after collecting all Case Record Form
Frequency of changes in ambulant treatment according to the acceptance of the program. | up to 12 months
  after collecting all Case Record Form
Frequency of newly occurred symptomatic acute cardiac events according to the acceptance of the program. | up to 12 months
  after collecting all Case Record Form
Frequency of resource use according to the acceptance of the program. | up to 12 months
  after collecting all Case Record Form

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Brasch, Prof. Dr., Study Director — AstraZeneca Germany; Franz Goss, Dr. med., Principal Investigator — 80331 Munich, Germany
Locations (45):
- Germany (45):
  - Research Site, Arnstadt
  - Research Site, Augsburg
  - Research Site, Bad Soden
  - Research Site, Berlin
  - Research Site, Berlin-Helersdorf
  - Research Site, Berlin-Humbold
  - Research Site, Berlin-Pankow
  - Research Site, Berlin-Spandau
  - Research Site, Bonn
  - Research Site, Buchholz
  - Research Site, Chemnitz
  - Research Site, Coburg
  - Research Site, Cologne
  - Research Site, Coswig
  - Research Site, Cottbus
  - Research Site, Dessau
  - Research Site, Dinslaken
  - Research Site, Düsseldorf
  - Research Site, Flensburg
  - Research Site, Frankfurt
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Hilden
  - Research Site, Höchberg
  - Research Site, Höxter
  - Research Site, Karlstadt am Main
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Lichtenberg
  - Research Site, Lippstadt
  - Research Site, Loerrach
  - Research Site, Lünen
  - Research Site, Magdeburg
  - Research Site, Merseburg
  - Research Site, Neukölln
  - Research Site, Nordhausen
  - Research Site, Querfurt
  - Research Site, Regensburg
  - Research Site, Stralsund
  - Research Site, Templin
  - Research Site, Ulm
  - Research Site, Ulm Donau
  - Research Site, Wesel
  - Research Site, Wilster
  - Research Site, Würzburg